CLINICAL TRIAL: NCT00086255
Title: Tiagabine for the Treatment of Cocaine Dependence
Brief Title: Tiagabine for the Treatment of Cocaine Dependence - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Cincinnati (Other)
Responsible Party: Liza Gorgon / Clinical Trials Specialist, NIDA
Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-CTO-0012-1
Record Dates: First submitted 2004-06-29; First posted 2004-06-30 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2008-08

CONDITIONS: Cocaine-Related Disorders
Keywords: cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Tiagabine

INTERVENTIONS:
Drug: Tiagabine

SUMMARY:
The purpose of this study is to assess tiagabine for the treatment of cocaine dependence.

DETAILED DESCRIPTION:
To assess the efficacy and safety of tiagabine in reducing cocaine use in subjects with cocaine dependence. It is hypothesized that tiagabine treatment, compared to placebo, will be associated with fewer days of cocaine use as assessed by self-report confirmed with urine assays for benzoylecgonine (BE). This is a double-blind, placebo-controlled, parallel-group design study, in which, after screening and a 2-week baseline assessment period, subjects will be equally randomly assigned to 1 of 2 treatment groups, tiagabine or matched placebo.

ELIGIBILITY:
Inclusion Criteria:

Must be at least 18 years of age and be seeking treatment for cocaine dependence. Have the ability to understand, and having understood, provide written informed consent. If female, agree to use a method of birth control as indicated by the clinician. Please contact the participating site in your area for more information.

Exclusion Criteria:

Please contact the participating site in your area for more information.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140
Dates: Start 2002-10; Study Completion 2004-06

PRIMARY OUTCOMES:
Drug use
Cocaine use
Addiction severity
Clinical improvement

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Somoza, M.D., Ph.D., Principal Investigator — Cincinnati VA Medical Center
Locations (4):
- United States (4):
  - Boston University Medical Center, Boston, Massachusetts
  - Cincinnati VA Medical Center, Cincinnati, Ohio
  - Dayton VA Medical Center, Dayton, Ohio
  - University of Texas Hlth Sci Ctr Houston, Houston, Texas

REFERENCES:
- [Derived] Winhusen TM, Somoza EC, Lewis DF, Kropp F, Theobald J, Elkashef A. An Evaluation of Substance Abuse Treatment and HIV Education on Safe Sex Practices in Cocaine Dependent Individuals. ISRN Addict. 2014 Mar 4;2014:912863. doi: 10.1155/2014/912863. eCollection 2014. PMID 25938124